CLINICAL TRIAL: NCT03579420
Title: Efficacy of a Brief Group Program Versus a Longer Structured Program for Therapeutic Education of Patients With Type 2 Diabetes.
Brief Title: Efficacy of a Brief Lifestyle Intervention in Type 2 Diabetes, Compared With a Longer Group Educational Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bPEGT2
Record Dates: First submitted 2018-06-01; First posted 2018-07-06 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief lifestyle program (Experimental): 3-session lifestyle group intervention program focussed on physical activity and eating habits, using interactive methods and a behavioral approach
  Interventions: Behavioral: Brief lifestyle program
- Traditional lifestyle longer program (Active Comparator): 6-session lifestyle group intervention program focussed on physical activity and eating habits, using traditional lessons and interactive methods
  Interventions: Behavioral: Conventional lifestyle program

INTERVENTIONS:
Behavioral: Brief lifestyle program — 3-session program for modification of lifestyle habits (exercise and diet)
  Arms: Brief lifestyle program
Behavioral: Conventional lifestyle program — 6-session program for modification of lifestyle habits (exercise and diet)
  Arms: Traditional lifestyle longer program

SUMMARY:
The study will compare two different programs for lifestyle intervention in type 2 diabetes:

1. A brief group program, with three weekly sessions
2. A longer group program, with six weekly sessions, which has been routinely used for the management of type 2 diabetic patients in this hospital for several years.

The aim is that of demonstrating the non-inferiority of the new brief, and more sustainable, program, in comparison with the more traditional approach.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c between 48 and 75 mmol/mol

Exclusion Criteria:

* Axis I Mental Disorders
* Heart failure (NYHA Class III or IV)
* Foot ulcers or lower limb amputations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c at 6 months | 6 months
Treatment success at 6 months | 6 months
  HbA1c within predefined target without any increase in pharmacological therapy

SECONDARY OUTCOMES:
Treatment success at 24 months | 24 months
  HbA1c within predefined target without any increase in pharmacological therapy
HbA1c at 24 months | 24 months
MEditerranean DIet adherence LITErature-based (MEDI-LITE) questionnaire scores | 24 months
  14-item questionnaire with scores ranging from 0 (low adherence) to 18 (high adherence)
International Physical Activity Questionnaire-Short Form (IPAQ-SF) scores | 24 months
  7-item questionnaire with scores ranging from 0 (no activity) to 7 (high activity)
Well-being Enquiry in Diabetics (WED) questionnaire total score | 24 months
  50-item questionnaire measuring diabetes-specific health-related quality of life, with scores ranging from 0 (low) to 50 (high). Only total score will be used in analysis 1. Mannucci E, et al., Diabetes Nutr Metab 9: 89-102, 1996).
Body Mass Index | 6 months
Waist circumference | 6 months
Body Mass Index | 24 months
Waist circumference | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetologia AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No